CLINICAL TRIAL: NCT00392314
Title: Phase 2 Study.Tailored Therapy for Hodgkin Lymphoma Based on Predefined Risk Factors and Early Interim PET/CT for Response Assessment and Further Therapy Decisions.
Brief Title: Tailored Therapy for Hodgkin Lymphoma Using Early Interim Therapy PET for Therapy Decision.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Collaborators: Hadassah Medical Organization (Other); Rabin Medical Center (Other)
Responsible Party: Principal Investigator, e_dann, Eldad J Dann assoc Prof of Hematology (Clinical), director of blood bank and aphaeresis unit RAMBAM health care campus Haifa Israel, Rambam Health Care Campus
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ISRA2432_CTIL
Record Dates: First submitted 2006-10-25; First posted 2006-10-26 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Hodgkin Lymphoma
Keywords: hodgkin lymphoma; PET/CT; Therapy
MeSH Terms: conditions — Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Early favorable (Experimental): patients with early favorable disease Ia IIA will have a PET/CT following 2 cycles of ABVD
  Interventions: Other: PET/CT post 2 cycles of chemotherapy
- Early Unfavorable (Experimental): Patients with early favorable disease Ia or IIa with risk factors :large mediastinal mass extra nodal disease elevated esr, three or more involved areas, age equal or >50 , lymphocytic depleted or mixed cellularity
  Interventions: Other: PET/CT post 2 cycles of chemotherapy
- advanced disease (Experimental): patients with advanced disease low IPS score 0-2 will start chemotherapy with ABVD for 2 cycles followed by PET/CT further therapy will be given according to PET/CT results
  Interventions: Other: PET/CT post 2 cycles of chemotherapy
- advanced disease IPS 3-7 (Experimental): Patients with advanced disease IPS score 3-7 will start chemotherapy with escalated beacopp. following 2 cycles PET/CT will be carried out and according to results further chemotherapy will be given
  Interventions: Other: PET/CT post 2 cycles of chemotherapy

INTERVENTIONS:
Other: PET/CT post 2 cycles of chemotherapy — sintigraphy with PET/CT following 2 cycles of chemotherapy on day 12-14 following chemotherapy
  Other Names: F18 deoxyglucose scintigraphy

SUMMARY:
Recently published studies demonstrated very high event free survival for patients with a normal interim PET/CT and a high hazard ratio for progression of an interim positive (pathological)study. These findings strongly support the integration of interim PET as a decision point for adjustment of chemotherapy.This study use the minimal therapy considered safe according to the predefined risk factors for patients with interim negative PET. Those with pathologic interim study considered as higher risk patients will have dose escalation of therapy.remission rate ,event free survival and overall survival will be evaluated.

DETAILED DESCRIPTION:
study aim is to tailor the therapy in order to administer the lowest cumulative dose of therapy yet considered safe in order to reduce both early and late therapy related complications.

patients will be divided according to risk factors to sub groups of early favorable, early unfavorable, advanced disease with score less then 3 points or higher then 3 points.

Early Interim PET will be carried out Further therapy will be based on the study results.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin lymphoma patients
* age 18-60 for those with early disease and advanced disease with score less then 3
* age 18-60 years for patients with advanced disease score 3 or higher classical Hodgkin lymphoma
* WBC more then 3500
* platelets more then 100000
* creatinin less then 2.0 mg
* bilirubin less then 2.0 mg
* absolute neutrophil count more then 1000 unless bone marrow involvement If marrow involve, patient with lower count but ANC of 1000 may be included.

Exclusion Criteria:

* Positive serology for HIV
* bilirubin more then 2 mg/dl
* creatinin more then 2 mg/dl
* lactating woman or pregnant
* patient older then 60 years with high risk disease of score 3 or more

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 365 (Actual)
Dates: Start 2006-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Event Free survival in various risk groups of patients | five years
Event Free Survival | 5 years

SECONDARY OUTCOMES:
overall survival5 years | 5 years
event free survival 5 years | five years
Disease free survival 5 years | five years

CONTACTS AND LOCATIONS:
Overall Officials: Eldad J Dann, MD, Study Chair — RABMAM medical center ,Haifa Israel , Rappapport school of medicine Technion Israel technical Institute Haifa Israel
Locations (1):
- RAMBAM health care campus, Haifa, Israel